CLINICAL TRIAL: NCT04640025
Title: A Phase 2, Open-Label, Multicenter, Rollover Study to Provide Continued Treatment for Participants Previously Enrolled in Studies of Itacitinib (INCB039110)
Brief Title: A Rollover Study to Provide Continued Treatment for Participants Previously Enrolled in Studies of Itacitinib
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INCB 39110-801; 2022-501661-47-00 (Registry Identifier: EU CT Number); 2020-002134-32 (EudraCT Number)
Expanded Access: NCT05561985 (Available)
Record Dates: First submitted 2020-11-18; First posted 2020-11-23 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Myelofibrosis; Postlung Transplant (Bronchiolitis Obliterans); Chronic Graft Versus Host Disease
Keywords: itacitinib; INCB39110
MeSH Terms: conditions — Primary Myelofibrosis; Bronchiolitis Obliterans; Bronchiolitis Obliterans Syndrome | interventions — itacitinib; INCB039110

STUDY DESIGN:
Intervention Model Description: Individual patients will continue to be treated with itacitinib in accordance with the parent study under which they were enrolled.
Masking Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- itacitinib (Experimental): Participants will receive treatment with itacitinib as per the treatment dose and schedule they received in the study in which they were originally enrolled. Participants who are receiving ruxolitinib under parent protocol INCB39110-209 may continue to receive it as described in that protocol.
  Interventions: Drug: itacitinib

INTERVENTIONS:
Drug: itacitinib — Participants will self-administer itacitinib orally using intact tablets with water and without regard to food.
  Other Names: INCB039110

SUMMARY:
This is a mutli-center open-label study to provide continued supply of itacitinib to participants from the following Incyte-sponsored studies of itacitinib: INCB39110-209, INCB39110-213, INCB39110-214, INCB39110-230, and 39110-309. Eligible participants will receive treatment with itacitinib as per the treatment dose and schedule they received in the study in which they were originally enrolled. The original study is referred to as the "parent protocol".

Participants who receive itacitinib in this study may continue treatment as long as the regimen is tolerated, the participant is deriving clinical benefit (in the opinion of the investigator), and the participant does not meet discontinuation criteria.

ELIGIBILITY:
Inclusion Criteria:

* Currently enrolled and receiving treatment in an Incyte-sponsored itacitinib (INCB39110)-based clinical study (parent Protocol).
* Currently tolerating treatment as defined by the parent Protocol.
* Currently receiving clinical benefit from itacitinib-based treatment, as determined by the investigator.
* Has demonstrated compliance, as assessed by the investigator, with the parent protocol requirements.
* Willingness and ability to comply with scheduled visits, treatment plans, and any other study procedures indicated in this Protocol.
* Willingness to avoid pregnancy or fathering children..
* Ability to comprehend and willingness to sign an ICF.

Exclusion Criteria:

* Able to access itacitinib therapy commercially.
* Participants with an uncontrolled intercurrent illness or any concurrent condition that, in the investigator's opinion, would jeopardize the safety of the participant or compliance with the Protocol.
* Pregnant or breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2026-06-22 (Estimated); Study Completion 2026-06-22 (Estimated)

PRIMARY OUTCOMES:
Treatment Emergent Adverse Events (TEAE's) | 3 years
  Adverse events reported for the first time or worsening of a pre-existing event after first dose of study drug/treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Lance Leopold, MD, Study Director — Incyte Corporation
Locations (21):
- United States (8):
  - City of Hope National Medical Center, Duarte, California
  - Anschutz Cancer Pavilion-University of Colorado, Aurora, Colorado
  - Parkview Cancer Institute, Fort Wayne, Indiana
  - Cleveland Clinic, Cleveland, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Temple University Department of Thoracic Medicine and Surgery, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Texas Oncology San Antonio, San Antonio, Texas
- Ordensklinikum Linz Gmbh Elisabethinen, Linz, Austria
- Universitaire Ziekenhuis Leuven - Gasthuisberg, Leuven, Belgium
- Providence Health, Vancouver, British Columbia, Canada
- Germany (3):
  - Universitatsklinikum Halle (Saale), Halle
  - University Medical Centre Hamburg-Eppendorf Centre of Oncology, Hamburg
  - University Hospital Mannheim, Mannheim
- University Hospital of West Attica - Attikon, Chaïdári, Greece
- Hadassah Hebrew University Medical Center Ein Karem Hadassah, Jerusalem, Israel
- Italy (3):
  - Azienda Policlinico Vittorio Emanuele, Catania
  - Azienda Ospedaliera Bianchi-Melacrino-Morelli Ospedali Riuniti, Reggio Calabria
  - Aou San Giovanni Di Dio E Ruggi, Salerno
- Spain (2):
  - Hospital Universitario Virgen de Las Nieves, Granada
  - Hospital Universitario Ramon Y Cajal, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency

REFERENCES:
- See also: A Rollover Study to Provide Continued Treatment for Participants Previously Enrolled in Studies of Itacitinib — https://incyteclinicaltrials.com/studies/incb-39110-801